CLINICAL TRIAL: NCT07263828
Title: The Effect of a Breathing Meditation Program on Perceived Stress, Sense of Integrity, and Quality of Life in the Elderly: A Randomized Controlled Study
Brief Title: Breath Meditation on the Older People
Acronym: MEDITATION
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, DİLEK YILDIRIM, Associate Professor, Istanbul Aydın University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Breath Meditation on the Older
Record Dates: First submitted 2025-11-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: Individuals Over 65 Years of Age
Keywords: Mindfulness; Psychological Stress; Nursing, Breathing Meditation; Breathing Exercises; Quality of Life; Older
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional (Experimental): Individuals in the experimental group were given a 15-minute breathing meditation session every day for 10 days.
  Interventions: Other: breathing meditation
- Control (No Intervention): No-application group

INTERVENTIONS:
Other: breathing meditation — Individuals in the experimental group were given a 15-minute breathing meditation session every day for 10 days.
  Arms: Interventional

SUMMARY:
A decrease in physical activity during old age leads to a decline in quality of life and life satisfaction. Increased stress and anxiety levels during this period negatively affect individuals' mood and reduce their quality of life. Individuals with a strong sense of coherence cope more effectively with stress and maintain a higher quality of life. Breathing meditation is a side-effect-free and easily applicable method that reduces the effects of stress by increasing individual awareness. Mindfulness-based breathing practices contribute to mental calmness and a healthier coping with stress. Experimental studies evaluating the effects of breathing meditation on stress, sense of coherence, and quality of life in older individuals are limited in the literature. This study aimed to determine the effects of a breathing meditation program on perceived stress, sense of coherence, and quality of life in older individuals.

The study was conducted with a randomized controlled experimental design between October 2024 and September 2025 with 128 participants (63 in the experimental group and 65 in the control group). Data were collected using the Participant Information Form, the Perceived Stress Scale (PSS), the Sense of Personal Integrity Scale (SWI), and the Quality of Life Scale for the Elderly (WHOQOL-OLD). Individuals in the experimental group received a 15-minute breathing meditation session daily for 10 days. The control group received no intervention. The scales were administered as a pretest and a posttest after day 15 in both groups. Data were analyzed using SPSS software; independent and dependent sample t-tests, chi-square tests, and descriptive statistics were used, with a significance level of p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 65 years and above,
* who volunteered to participate,
* had no communication difficulties,
* had not previously received any training or practice related to relaxation, breathing, or stress management.

Exclusion Criteria:

* Having received any training or practice in relaxation, breathing or stress management before.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Participant Information Form | Baseline- first day
  The Participant Information Form was developed by the researchers in line with the literature and included sociodemographic characteristics such as age, gender, marital status, educational level, and living situation
Perceived Stress Scale | Baseline (First day)
  The scale consists of 14 items rated on a 5-point Likert scale ranging from 0 ("never") to 4 ("very often"), with higher scores indicating higher levels of perceived stress. Negatively worded items are reverse-scored, and the total score ranges from 0 to 56.
The Sense of Coherence Scale | Baseline (First day)
  The scale consists of 13 items rated on a 7-point Likert scale, and higher scores indicate a stronger sense of coherence. The SOC captures how individuals understand and respond to life events, their perceived ability to manage challenges, and the meaningfulness they attribute to life experiences.
WHOQOL-OLD (World Health Organization Quality of Life - Older Adults Module | Baseline (First day)
  Quality of life was evaluated using the WHOQOL-OLD scale, developed by the World Health Organization for older adults. The scale includes 24 items covering six domains: sensory abilities, autonomy, past, present, and future activities, social participation, death and dying, and intimacy. Items are scored on a 5-point Likert scale, with higher scores indicating better quality of life.
Perceived Stress Scale | Post test - Fifteenth day
  The scale consists of 14 items rated on a 5-point Likert scale ranging from 0 ("never") to 4 ("very often"), with higher scores indicating higher levels of perceived stress. Negatively worded items are reverse-scored, and the total score ranges from 0 to 56.
The Sense of Coherence Scale | Post test - Fifteenth day
  The scale consists of 13 items rated on a 7-point Likert scale, and higher scores indicate a stronger sense of coherence. The SOC captures how individuals understand and respond to life events, their perceived ability to manage challenges, and the meaningfulness they attribute to life experiences.
WHOQOL-OLD (World Health Organization Quality of Life - Older Adults Module | Post test - Fifteenth day
  Quality of life was evaluated using the WHOQOL-OLD scale, developed by the World Health Organization for older adults. The scale includes 24 items covering six domains: sensory abilities, autonomy, past, present, and future activities, social participation, death and dying, and intimacy. Items are scored on a 5-point Likert scale, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sinop University, Sinop, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided